CLINICAL TRIAL: NCT01011478
Title: Statin Polyp Prevention Trial in Patients With Resected Colon Cancer
Brief Title: Rosuvastatin in Treating Patients With Stage I or Stage II Colon Cancer That Was Removed By Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSABP-P-5; NSABP P-5; NCI-2011-09183 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer; Precancerous Condition
Keywords: adenomatous polyp; stage I colon cancer; stage II colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Adenomatous Polyps; Colonic Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: placebo (Placebo Comparator): Patients receive oral placebo once daily for 5 years.
  Interventions: Other: placebo
- Group 2: rosuvastatin (Experimental): Patients receive oral rosuvastatin once daily for 5 years.
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin
  Other Names: Crestor
  Arms: Group 2: rosuvastatin
Other: placebo
  Arms: Group 1: placebo

SUMMARY:
RATIONALE: Rosuvastatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving rosuvastatin after surgery may kill any tumor cells that remain after surgery. It may also keep polyps from forming or colon cancer from coming back. It is not yet known whether rosuvastatin is more effective than a placebo in treating colon cancer that was removed by surgery.

PURPOSE: This randomized phase III trial is studying rosuvastatin to see how well it works compared with placebo in treating patients with stage I or stage II colon cancer that was removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the effect of rosuvastatin vs placebo on the 5-year occurrence of adenomatous polyps of the colon or rectum, metachronous colorectal carcinoma, or colon cancer recurrence (APMC+R) in patients with resected stage I or II colon cancer.

Secondary

* To determine whether the effect of rosuvastatin vs placebo is of the same magnitude in patients taking aspirin (regardless of dose) compared to patients not taking aspirin.
* To determine whether taking aspirin (regardless of dose) vs no aspirin will decrease the occurrence or APMC+R and, if there is an effect, to explore the relationship to dose.
* To determine the effect of rosuvastatin in patients with familial colorectal cancer.
* To determine the effect of rosuvastatin in patients with microsatellite unstable tumors (i.e., tumors displaying loss of MLH1 or MSH2 expression by IHC).
* To determine the relationship between rosuvastatin therapy and features of colorectal adenomas as well as the size and number of colorectal adenomas.
* To compare the time to APMC+R in patients treated with rosuvastatin vs placebo.
* To compare the disease-free survival of patients treated with rosuvastatin vs placebo.
* To compare the overall survival of patients treated with rosuvastatin vs placebo.
* To compare the rate of recurrence of colon cancer in patients treated with rosuvastatin vs placebo.
* To compare the rate of second non-colorectal primary cancers in patients treated with rosuvastatin vs placebo.
* To determine the effect of rosuvastatin on health-related quality of life, global quality of life, and self-reported symptoms.
* To compare the incidence and severity of adverse events associated with rosuvastatin vs placebo.
* To assess relevant tumor and blood markers that may affect the metabolism, activity, or effect of the study drugs, such as HMG-CoA reductase, UGT1A6, P450-2C9, PTGS2 (COX-2), and other possible markers.

OUTLINE: This is a multicenter study. Patients are stratified according to family history of a first-degree relative with colorectal cancer (yes vs no), intended aspirin dose (none vs 81 mg vs 325 mg), and adjuvant therapy for colon cancer (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Group 1: Patients receive oral placebo once daily for 5 years.
* Group 2: Patients receive oral rosuvastatin once daily for 5 years.

Patients may complete a quality-of-life questionnaire at baseline and at 6, 12, 36, 60, and 84 months.

Tumor tissue, serum, and blood samples may be collected periodically for biomarker and other analyses.

After completion of study treatment, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria

* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must have the ability to swallow oral medication.
* Patients must have resected adenocarcinoma of the colon staged as American Joint Committee on Cancer (AJCC) Stage 0, I, II, or III.
* Patients must have had surgical resection of the colon adenocarcinoma with curative intent within 1 year prior to randomization. (Laparoscopically-assisted colectomy is permitted.)
* Patients must have completed any adjuvant therapy prior to randomization.
* Patients who are taking cardioprotective low-dose aspirin at study entry must not have clinically significant toxicity, as determined by the investigator, that precludes continuation of aspirin, and the patient must be willing to continue aspirin therapy (81 mg or 325 mg) throughout study therapy.
* Colonoscopy requirements within 180 days prior to randomization:
* The patient must have either undergone a preoperative or postoperative documented colonoscopy to the cecum (or small bowel anastomosis) with adequate bowel preparation.
* All observed polyps must have been removed. (Polyps can be removed during colonoscopy or surgery performed prior to randomization.)
* Postoperative serum creatinine performed within 90 days prior to randomization must be less than or equal to 1.5 x upper limit of normal (ULN) for the lab.
* The following criteria for evidence of adequate hepatic function based on postoperative testing performed within 90 days prior to randomization must be met: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) less than or equal to 3.0 x ULN for the lab, and Total bilirubin less than or equal to 1.5 x ULN for the lab

Exclusion Criteria

* Tumor with the distal border located less than 12 cm from the anal verge.
* Total colectomy or total proctocolectomy.
* Classic Familial Adenomatous Polyposis, Attenuated Familial Adenomatous Polyposis (i.e., 20 or more adenomas, either synchronous or metachronous), or Hereditary Nonpolyposis Colorectal Cancer (Lynch Syndrome).
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease significantly affecting gastrointestinal function.
* History of documented upper GI bleeding or upper GI ulcerative disease.
* Statin use within 30 days prior to randomization.
* Hyperlipidemia with clinical indication for statin therapy or other prescribed medication. Determination of acceptable fasting lipid values, within 90 days prior to randomization, should be in accordance with current dyslipidemia management guidelines.
* Unwillingness to discontinue chronic use of nonsteroidal antiinflammatory drugs (NSAIDs) (other than cardioprotective low-dose aspirin 81 mg or 325 mg) prior to randomization.
* Anticipated need for chronic use of NSAIDs (other than cardioprotective low-dose aspirin 81 mg or 325 mg).
* Inadequately treated hypothyroidism, as determined by the investigator.
* History of myopathy or rhabdomyolysis.
* Hypersensitivity or intolerance to statins.
* Chronic drug therapy with cyclosporine, coumarin anticoagulants, gemfibrozil, some other lipid-lowering therapies (fibrates or niacin), lopinavir/ritonavir, or drugs (such as ketoconazole, spironolactone, or cimetidine) that lower levels or activity of steroid hormones.
* Pregnancy or lactation at the time of study entry. (Pregnancy testing must be performed within 14 days prior to randomization according to institutional standards for women of childbearing potential.)
* Previous malignancies unless the patient has been disease-free for 5 or more years prior to randomization and is deemed by the physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: all in situ cancers and basal cell and squamous cell carcinoma of the skin.
* Other non-malignant systemic disease that would preclude a patient from receiving rosuvastatin or would prevent prolonged follow-up.
* Administration of any investigational agent within 30 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (587):
- United States (584):
  - Regional Medical Center, Anniston, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Little Rock, Arkansas
  - Kaiser Permanente Medical Center - Anaheim/Orange County, Anaheim, California
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente Medical Center - Baldwin Park, Baldwin Park, California
  - Kaiser Permanente Medical Center - Bellflower, Bellflower, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente Medical Center - Fontana, Fontana, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Kaiser Permanente Medical Center - Harbor City, Harbor City, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente - Irvine, Irvine, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Kaiser Foundation Hospital - West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Epic Care - Oakland, Oakland, California
  - Kaiser Permanente - Ontario Vineyard Medical Offices and Ambulatory SurgiCenter, Ontario, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Kaiser Permanente Medical Group, Panorama City, California
  - Lucy Curci Cancer Center at Eisenhower Memorial Hospital and Medical Center, Rancho Mirage, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Riverside, Riverside, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Kaiser Permanente Medical Cener - Woodland Hills, Woodland Hills, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Bendheim Cancer Center at Greenwich Hospital, Greenwich, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Kent General Hospital, Dover, Delaware
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Kaiser Permanente at Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - CHRISTUS Cabrini Cancer Center, Alexandria, Louisiana
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Mercy Hospital, Portland, Maine
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Kaiser Permanente at Woodlawn Medical Center, Baltimore, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Kaiser Permanente - Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Southcoast Center for Cancer Care, Fairhaven, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Regional Cancer Center, Pennington, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Celilo Cancer Center at Mid-Columbia Medical Center, The Dalles, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Kaiser Permanente Medical Center - Fair Oaks, Fairfax, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Olympic Medical Cancer Center, Sequim, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - St. Mary Regional Cancer Center at St. Mary Medical Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - United Hospital Center, Clarksburg, West Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
- Canada (3):
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec

REFERENCES:
- [Result] Boman BM, Bandos H, Wickerham DL, et al.: Statin polyp prevention trial in patients with resected colon cancer: NSABP protocol P-5. [Abstract] J Clin Oncol 30 (Suppl 15): A-TPS1615, 2012.

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Placebo: Patients receive oral placebo once daily for 5 years.
  placebo
- Group 2: Rosuvastatin: Patients receive oral rosuvastatin once daily for 5 years.
  rosuvastatin
Period: Overall Study
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Started | 204 | 202
Completed | 192 | 195
Not Completed | 12 | 7
Not completed — No follow up data | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
- Rosuvastatin: Rosuvastatin
- Total: Total of all reporting groups
Arm/Group | Placebo | Rosuvastatin | Total
Number analyzed (Participants) | 204 | 202 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.3) | 58 (10.9) | 58 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 108 | 221
  Male | 91 | 94 | 185

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of ≥ 1 Adenomatous Polyp of the Colon or Rectum, Metachronous Colorectal Carcinoma, or Colon Cancer Recurrence (APMC+R)
Description: Percentage of patients with occurrence of APMC+R event. APMC+R events include at least one adenomatous polyp of the colon or rectum, metachronous colorectal carcinoma, or colon cancer recurrence
Time Frame: Up to 4.8 years
Population: NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Number; unit: percentage of patients
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 192 | 195
percentage of patients | 25.0 | 28.2

2. Secondary Outcome: Size of Colorectal Adenomas, Including Advanced Adenomas
Description: The histologic size (diameter of adenoma into the wall of the colon; as per AJCC staging) of the largest adenoma among patients who have at least one adenoma detected. If histologic size was not available, the endoscopic size was provided.
Time Frame: Up to 4.8 years
Population: Patients who have at least one adenoma detected. NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Median (Inter-Quartile Range); unit: centimeters
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 46 | 50
centimeters | 0.4 [0.3 to 0.7] | 0.4 [0.3 to 0.55]

3. Secondary Outcome: Disease-free Survival
Description: Number of patients with DFS event (colon cancer recurrence, second primary cancer, or death from any cause)
Time Frame: Up to 4.8 years
Population: NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Number; unit: participants with DFS event
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 192 | 195
participants with DFS event | 17 | 21

4. Secondary Outcome: Overall Survival (OS)
Description: Number of patients with the OS event (death from any cause)
Time Frame: Up to 4.8 years
Population: NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Number; unit: participants with OS event
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 192 | 195
participants with OS event | 1 | 4

5. Secondary Outcome: Recurrence-free Interval (RFI)
Description: Number of patients with the RFI event (First recurrence of colon cancer)
Time Frame: Up to 4.8 years
Population: NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Number; unit: participants with RFI event
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 192 | 195
participants with RFI event | 12 | 14

6. Secondary Outcome: Second Non-colorectal Primary Cancer-free Interval
Description: Number of patients with the first occurrence of non-colorectal primary cancer
Time Frame: Up to 4.8 years
Population: NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Number; unit: participants non-colorectal primary cx
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 192 | 195
participants non-colorectal primary cx | 4 | 7

7. Secondary Outcome: Behavioral and Health Outcomes as Measured by SF-12 Component Scores, Global Quality-of-life Scale, and Symptom Checklist
Description: Global Quality-of-life Scale score, ranges from 0 (worst imaginable health status) to 10 (best imaginable health status.
Time Frame: 12-month time point
Population: Patients who have submitted a 12 months QOL assessment. NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 70 | 62
score on a scale | 8.0 [7 to 9] | 8.0 [8 to 9]

8. Secondary Outcome: Toxicity Assessed by Adverse Events
Description: Percentage of patients with at least one grade 2 or higher adverse event reported.
Time Frame: Up to 4.8 years
Population: Patients with available adverse event information. NOTE: No conclusions should be drawn due to insufficient number of patients randomized to the study.
Measure: Number; unit: percentage of patients
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 191 | 196
percentage of patients | 41.4 | 45.4

9. Secondary Outcome: Measurements of Relevant Tumor and Blood Markers
Description: This study terminated early. Data on samples was not collected, the relevant analyses were not performed.
Time Frame: At randomization
Population: Data on tumors and blood markers were not collected.
Arm/Group | Group 1: Placebo | Group 2: Rosuvastatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Placebo | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 17/191 | 14/196
Other Adverse Events (participants affected / at risk) | 28/191 | 34/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=191) | Rosuvastatin (N=196)
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 3
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 1 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=191) | Rosuvastatin (N=196)
Abdominal pain (Gastrointestinal disorders) | 7 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 14

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less